## **Analysis Plan**

Official Title: Veterans Justice Reentry (Post-Incarceration) (QUE 15-284)

Brief Title: Improving Linkage to Health and Other Services for Veterans Leaving Incarceration (PIE)

ClinicalTrials.gov ID: NCT02964897

**Unique Protocol ID: QUX 16-012** 

Study Principal Investigator: D. Keith McInnes, ScD MS BA

Document date: September 7, 2021

## **Analysis Plan:**

## Improving Linkage to Health and Other Services for Veterans Leaving Incarceration (ID QUX 16-012)

We will enroll Veterans on a rolling basis as released from MA correctional facilities. We will use HOMES database to create a historical comparison group comprised of all Veterans released in MA in the two-year period directly preceding the start of the PIE intervention and who accessed VA Health Care for Reentry Veterans (HCRV) services.

Quantitatively, we will use HOMES and CDW to compare intervention and comparison Veterans with respect to their baseline demographic characteristics (age, gender, race, ethnicity, marital status, self-rated health) and our outcomes interest. Also for intervention Veterans we will have self-report diagnoses and utilization from baseline and 6-month follow up (including utilization of non-VA health care sources). We will compare rates of visits for primary care, outpatient MH treatment, outpatient SUD treatment, as well as missed opportunities (e.g. no shows) between intervention and comparison groups using t-tests and chi-square tests. For our secondary measures we will also compare intervention to comparison on ER and hospital use (episodes and # of days) during the 6-month reentry period.

Analysis involves two phases. First, we use descriptive statistics to summarize the volume and intensity of peer activities in support of the Post-Incarceration Engagement (PIE) intervention participants. Secondly, to examine access to and engagement in care outcomes, we compare our measures of linkages to VA health care following release between PIE participants and our historical comparison group. Specifically, we use bivariate tests (Chi-Square/Fisher Exact Tests and t-tests, as appropriate) to assess the relationship between participation in the PIE intervention and linkages with VA health care.

## Summary of key variables

- Demographics (age, gender, race, ethnicity, marital status, self-rated health)
- SUD diagnoses
- MH diagnoses
- Criminal offense
- Length of incarceration
- # of arrests
- Housing/homeless experience
- Major comorbidities (out of list of 10-12)
- Visits to primary care
- Visits to MH outpatient care
- Visits to SUD outpatient care
- ED encounters
- Inpatient hospitalizations
- No shows at the above appointments

All data will be stored on VINCI and all analysis will be conducted on VINCI